CLINICAL TRIAL: NCT05219370
Title: Treatment With Cannabis Oil Containing Canabidiol (CBD) Tetrahydrocannabinol (THC), Cannabidivarin (CBDV) or Cannabigerol (CBG) vs. Placebo of Persons Diagnosed With ADHD After Failure of Conventional Treatment
Brief Title: Treatment With Cannabis Oil Containing CBD, THC, CBDV or CBG vs. Placebo of Persons With ADHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in enrollment
Sponsor: Brlev Agricultural Crops Ltd (Industry)
Collaborators: Bio-Sciences Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0232-19-ASF
Record Dates: First submitted 2021-12-30; First posted 2022-02-02 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: ADHD; Hyperactivity; Attention Deficit
Keywords: medical cannabis
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: each participant will be randomized to one of the 4 arms and will receive the treatment for 32 days. Follow up till 6 weeks from starting
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the responsible pharmacist is un-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CBD rich (Experimental): Cannabis oil oral drops containing 95 mg/ml CBD; 5 mg/ml THC; 15 mg/ml CBDV ; no CBG, once daily Titration from 0.3 to 1.8 ml/day during 21 days
  Interventions: Drug: Cannabis oil
- CBG rich (Experimental): Cannabis oil oral drops containing no CBD; 5 mg/ml THC; no CBDV; 95 mg/ml CBG, once daily.
  Titration from 0.3 to 1.8 ml/day during 21 days
  Interventions: Drug: Cannabis oil
- CBD & CBG rich (Experimental): Cannabis oil oral drops containing 47.5 mg/ml CBD; 2.5 mg/ml THC; 7.5 mg/ml CBDV; 47.5 mg/ml CBG, once daily.
  Titration from 0.3 to 1.8 ml/day during 21 days
  Interventions: Drug: Cannabis oil
- placebo (Placebo Comparator): Placebo oil oral drops once daily. Titration from 0.3 to 1.8 ml/day during 21 days
  Interventions: Drug: Cannabis oil

INTERVENTIONS:
Drug: Cannabis oil — administration of different cannabis oil types as compared with placebo

SUMMARY:
ADHD is the most frequent neuro-developmental disorder in childhood and often continues into adolescence and adulthood.

Indicated drug treatments for ADHD fall into 2 categories: stimulants (such as methylphenidate and amphetamines) and non-stimulants (such as atomoxetine, guanfacine and clonidine) but some persons cannot tolerate their secondary effects or find them non-effective.

In the last decade, medical cannabis products have been researched as possible treatment for neurological and mental diseases such as: Post trauma disorder (PTD), autism (ASD), epilepsy, fibromyalgia (FM) and more.

Data on the effects of cannabidiol rich cannabis extract use for ADHD seems promising but is still limited. The aim of this study is to investigate if oral cannabinoids given to adults with ADHD affect the symptoms of the disorder.

The main objectives of the study are: 1) to characterize the effects of treatment with cannabis oil on symptoms of ADHD; 2) to compare safety and efficacy of cannabis oil products with different CBD,Cannabidivarin (CBDV), cannabigerol (CBG) and THC ratio; 3) and to measure endocannabinoids, THC and CBD and metabolites levels in the blood of the participants.

In this study, participants diagnosed with ADHD will be treated with canabidiol-rich cannabis oil and will follow up weekly during approx.1 month (the study period). Blood tests will be performed before and after treatment. Blood tests include blood count, blood chemistry, hormones profile, phyto- and endo- cannabinoids and their metabolites. Test of Variables of Attention test (TOVA) will be administrated before and after treatment

DETAILED DESCRIPTION:
Participants will be screened by study staff for ADHD diagnosis and failure of conventional treatment.

Participants passing the screening will undergo blood and urine tests, fill questionnaires, TOVA test and will be randomized to one of the 4 arms.

Participants will receive the drug, be instructed as per dose titration and as per danger of driving under drug influence.

Telephone follow up will take place weekly after 7 days from starting. Participants will guess to which arm the participant was allocated to after 2 weeks of treatment .

Participants will arrive for a last visit, fill questionnaires, do TOVA test and undergo blood and urine tests.

Participants will be contacted over the phone for a last time, after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged at least 18 y/o diagnosed with ADHD by Diagnostic and Statistical Manual of Mental Disorders (DSM)
* Participants with a lower than 0 TOVA score or with a higher than 0 score whom as per investigator opinion suffer from ADHD
* Participants who experienced treatment failure with more than one ADHD conventional drug
* Participants willing to attend all the visits in the trial.

Exclusion Criteria:

* Participants who were treated with benzodiazepines, antihistamines, etc, in the week that preceded the trial start.
* Participants suffering from neurologic or psychiatric diseases
* Participants suffering from malignant diseases
* Participants suffering from syndromes or metabolic diseases
* Participants with significant clinical diagnosis that can damage the trial unfolding. The investigator may include them after the end of the situation which prevented their previous inclusion.
* Participants breastfeeding, pregnant or not willing to use contraceptives.
* Participants that will not adhere to the protocol as per investigator opinion
* Participants who weight less than 45 kg or more than 120kg or with BMI greater than 30
* Participants participating in another clinical trial which includes drug treatment
* Participants receiving any treatment for ADHD
* Participants using drugs
* Participants using cannabis or products containing cannabinoids, including medical cannabis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy of cannabis oil on ADHD symptoms as per TOVA test | 30-35 days
  To assess if participants treated with cannabis oil show an improvement in TOVA scores
efficacy of cannabis oil on ADHD symptoms as per Conners questionnaire | 30-35 days
  To assess if participants treated with cannabis oil show an improvement in Conners score

SECONDARY OUTCOMES:
to assess side effects and their severity using questionnaire | 60 days
  To examine whether cannabis oil side effects are tolerable and transient
number of participants who dropped-out | 60 days
  to check whether drop out percentage is similar among groups

CONTACTS AND LOCATIONS:
Overall Officials: Mati Berkovitch, Principal Investigator — Shamir (Assaf Harofeh) Medical Center
Locations (1):
- Shamir (Assaf Harofeh) Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Statistical Analysis Plan to be shared
Supporting Information: Study Protocol, SAP
Time Frame: during all the trial
Access Criteria: interested colleagues

REFERENCES:
- [Result] Thomas R, Sanders S, Doust J, Beller E, Glasziou P. Prevalence of attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. Pediatrics. 2015 Apr;135(4):e994-1001. doi: 10.1542/peds.2014-3482. Epub 2015 Mar 2. PMID 25733754
- [Result] Cooper RE, Williams E, Seegobin S, Tye C, Kuntsi J, Asherson P. Cannabinoids in attention-deficit/hyperactivity disorder: A randomised-controlled trial. Eur Neuropsychopharmacol. 2017 Aug;27(8):795-808. doi: 10.1016/j.euroneuro.2017.05.005. Epub 2017 May 30. PMID 28576350

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05219370/Prot_SAP_000.pdf